CLINICAL TRIAL: NCT01932242
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of Repeat Administration of Intravenous ETI-204 in Adult Volunteers
Brief Title: Safety, Tolerability and PK of Repeat Administration of Intravenous ETI-204 in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elusys Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AH109
Record Dates: First submitted 2013-08-02; First posted 2013-08-30 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-01

CONDITIONS: Inhalational Anthrax
Keywords: anthrax, monoclonal antibody, ETI-204, safety, PK
MeSH Terms: conditions — Inhalation anthrax; Anthrax | interventions — obiltoxaximab

STUDY DESIGN:
Intervention Model Description: Seventy subjects will be randomized in a 1:1 ratio to one of the following two treatment sequences:
  * Sequence A: ETI-204 on Days 1 and 14 and placebo on Day 120
  * Sequence B: ETI-204 on Days 1 and 120 and placebo on Day 14
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study drug will be prepared by an unblinded pharmacist not involved with the conduct of the study. The pharmacist will assign the correct study drug (16 mg/kg ETI-204 or placebo) to each subject according to the randomization scheme.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): An intravenous dose of 16 mg/kg ETI-204 infused over 90 minutes on Days 1 and 14 and an intravenous dose of ETI-204-Placebo infused over 90 minutes on Day 120.
  Interventions: Biological: ETI-204; Other: Placebo
- Sequence B (Experimental): An intravenous dose of 16 mg/kg ETI-204 infused over 90 minutes on Days 1 and 120 and an intravenous dose of ETI-204-Placebo infused over 90 minutes on Day 14.
  Interventions: Biological: ETI-204; Other: Placebo

INTERVENTIONS:
Biological: ETI-204 — Monoclonal Antibody
Other: Placebo — Placebo for ETI-204

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and immunogenicity of repeat administration (two doses) of intravenous (IV) ETI-204.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, study in 70 healthy adult subjects. The total duration of the study for each subject will be approximately 220 days divided as follows:

* Screening: Days -28 to -2
* Three In-Unit Stays: Days -1 to 2; Days 13 to 15; and Days 119 to 121
* Out-of-Unit Visit Days: Day 8 (±2 days); Day 28 (±3 days); Day 43 (±3 days); Day 71 (±3 days); Day 85 (±3 days); Day 128 (±3 days); Day 134 (±3 days); Day 149 (±3 days); and Day 163 (±3 days)
* Final Visit: Day 191 (±3 days)

Subjects will be randomized in a 1:1 ratio to one of the following two treatment sequences:

* Sequence A: ETI-204 on Days 1 and 14 and placebo on Day 120
* Sequence B: ETI-204 on Days 1 and 120 and placebo on Day 14

Subjects who qualify for entry into the study following completion of the Screening visit will arrive at the clinical research unit (CRU) on Day -1. The next day, Day 1, qualified subjects will be randomized and will receive a single IV dose of ETI-204. Subjects will be pretreated with 50 mg oral diphenhydramine approximately 30 minutes prior to the start of the study drug infusion.

Subjects will be discharged from the CRU on Day 2, and will return to the CRU for an additional visit on Day 8.

Subjects will return to the CRU on Day 13 for their second in-unit stay. The next day, Day 14, subjects will be pretreated with 50 mg oral diphenhydramine and will receive study drug according to their randomized treatment assignment. Subjects will be discharged on Day 15 and will return to the CRU for four additional visits on Days 28 (±3 days), 43 (±3 days), 71 (±3 days), and 85 (±3 days).

Subjects will return to the CRU again on Day 119 for their third in-unit stay. On Day 120, subjects will be pretreated with 50 mg oral diphenhydramine and will receive study drug (either ETI 204 or placebo) according to their randomized treatment assignment. Subjects will be discharged on Day 121 and will return to the CRU for five additional visits on Days 128,134, 149, 163, and 191.

The first 20 subjects randomized and treated in the study will be dosed in groups of no more than 4 subjects/day. For the first 8 subjects, dosing of individual subjects on Day 14 and Day 120 will be separated by 30-60 minutes for safety monitoring. If no severe infusion reactions occur in any of the first 8 subjects at the time of the second dose, staggered dosing is not required for the remaining subjects receiving their second dose. Similarly, if no severe infusion reactions occur in any of the first 8 subjects at the time of the third dose, staggered dosing is not required for the remaining subjects receiving their third dose.

Enrollment of additional subjects will be paused until the first 20 subjects have received their second dose of study drug and a blinded review of the available clinical and laboratory AE data up to and including Day 15 is completed for the first 20 subjects. This review will be conducted by the Investigator in conjunction with the Clinical Trial Steering Committee and will focus on the possible development of new or more severe AEs with the Day 14 dose. If the outcome of this review is satisfactory, dosing of additional subjects will be permitted to continue in groups larger than 4 subjects. In the event that significant AEs are observed and unblinding should become necessary, it will be performed by an independent statistician who is not involved with the conduct of the study.

A second blinded safety review will be completed at least two weeks before any subject receives the third dose of study drug, (i.e. before any subject is dosed on Day 120). The Investigator in conjunction with the Clinical Trial Steering Committee will review all AEs seen to date in the study. This review will focus on AE data seen in association with the second infusion (Day14). If the outcome of this review is satisfactory, subjects may receive their third dose of study drug.

A third blinded safety review will be conducted after the initial cohort of 20 subjects has completed Day 121. No additional subjects should receive a third dose of study medication until the Investigator along with the Clinical Trial Steering Committee has completed a blinded safety review of the Day 120 and 121 clinical and laboratory AE data. This review will focus on the development of new or more severe AEs seen with repeat dosing. If the outcome of this review is satisfactory, the remaining subjects may receive their third dose of study drug.

In the event that significant AEs are observed and unblinding becomes necessary it will be performed by an independent statistician who is not involved with the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males ≥ 18 years of age
2. All females, regardless of childbearing potential, must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test at Screening and Day -1
3. Females of childbearing potential (i.e., not postmenopausal or surgically sterile) must agree to practice abstinence or to use a medically accepted method of contraception from the time of Screening through 30 days after the final study visit. Acceptable methods of contraception include diaphragm with spermicide; sponge with spermicide; condom with spermicide; or intrauterine device with condom or spermicide. The following contraceptive methods are acceptable only when used with a condom and spermicide: birth control pills, birth control patches, vaginal ring, hormone under the skin, or hormone injections
4. Postmenopausal females, defined as females who have had amenorrhea for at least 12 months either naturally or following cessation of all exogenous hormonal treatments, and have a follicle-stimulating hormone (FSH) level of > 40 mIU/mL at Screening
5. Females who have undergone surgical sterilization, including hysterectomy, bilateral oophorectomy, bilateral salpingectomy, tubal ligation, or tubal essure
6. Males must agree to practice abstinence or use a condom with spermicide and refrain from sperm donation during the study and for 30 days after the final study visit
7. Provide written informed consent
8. Willing to comply with study restrictions

Exclusion Criteria:

1. Pregnant or lactating woman
2. Clinically significant comorbidity that would interfere with completion of the study procedures or objectives or compromise the subject's safety
3. Seated systolic blood pressure (BP) ≥ 150 mmHg or ≤ 90 mmHg or diastolic BP ≥ 95 mmHg
4. Use of H1 receptor antagonists (i.e. antihistamines) within 5 days prior to Day 1
5. Evidence of drug or alcohol abuse as determined by the Investigator within 6 months of Day 1
6. Positive test result for drugs of abuse (with the exception of medically prescribed drugs) at Screening or on Day -1
7. Positive test for alcohol at Screening; exclusion is at the Investigator's discretion; subjects who test positive for alcohol at Day -1 are excluded from the study
8. Treatment with an investigational agent within 30 days or five half-lives of the investigational agent at Day 1 (whichever is longer)
9. Congenital or acquired immunodeficiency syndrome
10. Prior solid organ or bone marrow transplant
11. Positive test for Hepatitis B (surface antigen), Hepatitis C, or human immunodeficiency virus (HIV) at Screening
12. History of prior treatment for anthrax exposure or prior anthrax infection
13. Prior immunization with any approved or investigational anthrax vaccine or prior treatment with an approved or investigational anthrax treatment (i.e., ETI-204, raxibacumab, or anthrax immune globulin)
14. Military personnel deployed in 1990 or after, unless the subject can provide documentation demonstrating they have not previously received any approved or investigational anthrax vaccine
15. Use of systemic steroids, immunosuppressive agents, anticoagulants, or anti-arrhythmics within 1 year prior to Day 1. A single short course (i.e., less than 14 days) of systemic steroid therapy is allowed provided it concluded more than 6 months prior to Day 1
16. Donation or loss of > 500 mL of blood within 30 days or plasma within 7 days of Day 1
17. Prior stroke, epilepsy, relapsing or degenerative central nervous system disease, or relapsing or degenerative ocular disease
18. Myocardial infarction or acute coronary syndrome in the past 5 years, active angina pectoris, or heart failure (New York Heart Association scale > 1)
19. History of chronic liver disease
20. Calculated creatinine clearance (CrCl) of < 30 mL/min using the Cockcroft-Gault equation (see Section 5.1)
21. Any clinically significant abnormality, in the Investigator's opinion, on electrocardiogram (ECG) or clinical laboratory tests (hematology, clinical chemistry, or urinalysis) at Screening; Out of range results may be repeated to confirm.
22. History of allergic or hypersensitivity reactions to other therapeutic antibodies or immunoglobulins
23. History of any malignant neoplasm within the last 5 years, with the exception of adequately treated, localized or in situ non-melanoma carcinoma of the skin (e.g., basal cell carcinoma) or the cervix
24. Subjects who, in the opinion of the Investigator, are not suitable candidates for enrollment or who may not comply with the requirements of the study

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2014-04-19 (Actual); Study Completion 2014-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles, Inc.
Locations (2):
- United States (2):
  - Quintiles, Overland Park, Kansas
  - DaVita, Minneapolis, Minnesota

REFERENCES:
- [Derived] Nagy CF, Leach TS, Hoffman JH, Czech A, Carpenter SE, Guttendorf R. Pharmacokinetics and Tolerability of Obiltoxaximab: A Report of 5 Healthy Volunteer Studies. Clin Ther. 2016 Sep;38(9):2083-2097.e7. doi: 10.1016/j.clinthera.2016.07.170. Epub 2016 Aug 24. PMID 27568215

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: 16 mg/kg ETI-204 IV on Days 1 and 14 and Placebo on Day 120
  ETI-204: Monoclonal Antibody
  Placebo: Placebo for ETI-204
- Sequence B: 16 mg/kg ETI-204 IV on Days 1 and 120 and Placebo on Day 14
  ETI-204: Monoclonal Antibody
  Placebo: Placebo for ETI-204
Period: Overall Study
Arm/Group | Sequence A | Sequence B
Started | 35 | 35
Completed | 30 | 30
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (14.71) | 43.3 (16.76) | 43.1 (15.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 12 | 22
  White | 25 | 20 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Weight [Mean (Standard Deviation); unit: kg] | 83.19 (16.452) | 80.55 (16.886) | 81.87 (16.602)
Height [Mean (Standard Deviation); unit: cm] | 171.82 (10.623) | 172.46 (8.520) | 172.14 (9.564)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.23 (5.608) | 27.06 (5.275) | 27.65 (5.437)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety was assessed for all subjects in the safety population by collecting and monitoring vital signs, laboratory tests, ECGs, physical examinations, skin assessments, infusion site assessments and adverse events.
Time Frame: Up to 191 days or 221 days (30 days after the final study visit) for subjects with ongoing adverse events at the final study visit, for each arm.
Population: The safety population consisted of all subjects who received at least a partial dose of ETI 204 or placebo, whether prematurely withdrawn from the study or not
Measure: Count of Participants; unit: Participants
Groups:
- Sequence A: ETI-204 on Days 1 and 14 and placebo on Day 120
- Sequence B: ETI-204 on Days 1 and 120 and placebo on Day 14
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 35 | 35
Participants | 30 | 31

2. Secondary Outcome: Maximum Observed Plasma Concentration of ETI-204 (Cmax) After a Dose of 16 mg/kg on Day 1(Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: Blood samples were obtained and serum concentrations were determined using a validated enzyme-linked immunosorbent assay method with an assay range of 100 ng/mL to 5000 ng/mL.The PK parameter, Cmax, was derived from ETI-204 serum concentrations by sequence group and treatment period for the PK analysis population.
  Sequence A - there were insufficient serum concentration data to adequately characterize ETI 204 PK separately after each dose administration (Day 1 and Day 14), therefore it was treated as one 32 mg/kg dose split into two 16 mg/kg administrations. Sequence B was treated as 2 separate 16 mg/kg doses (Day 1 and Day 120).
  All 70 subjects who received ETI-204 were included in the PK population: 35 in Sequence A and 35 in Sequence B; however, the full complement of PK parameters could not be determined in all subjects.
Time Frame: On Days 1 and 14 predose, at the end of infusion, and 3 and 8 hours after the start of infusion, and on Days 2, 8, 15, 28, 43, 71, 85, 121, 128, 134, 149, 163, and 191.
Population: One subject in Sequence A was prematurely discontinued from the study by the investigator after the 1st dose of ETI-204 because of AEs. This subject did not receive the 2nd dose of ETI-204 on Day 14 and therefore all PK parameters from this subject were excluded from descriptive statistics.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 34 | 35
µg/mL | 506 (102) | 384 (103)

3. Secondary Outcome: Maximum Observed Plasma Concentration of ETI-204 (Cmax) After a Dose of 16 mg/kg on Day 120 (Sequence B)
Description: Blood samples were obtained and serum concentrations were determined using a validated enzyme-linked immunosorbent assay method with an assay range of 100 ng/mL to 5000 ng/mL.
  Sequence A - there were insufficient serum concentration data to adequately characterize ETI 204 PK separately after each dose administration (Day 1 and Day 14), therefore it was treated as one 32 mg/kg dose split into two 16 mg/kg administrations. Sequence B was treated as 2 separate 16 mg/kg doses (Day 1 and Day 120). All 70 subjects who received ETI-204 were included in the PK population: 35 in Sequence A and 35 in Sequence B; however, the full complement of PK parameters could not be determined in all subjects.
Time Frame: On Day 120 predose, at the end of infusion, and 3 and 8 hours after the start of infusion, and on Days 2, 8, 15, 28, 43, 71, 85, 121, 128, 134, 149, 163, and 191.
Population: Four subjects in Sequence B were excluded because the subjects did not receive the 2nd dose of ETI-204 16 m/kg on Day 120 (one due to AEs after the 1st dose, one withdrew consent due to conflict with work, one was lost to follow-up on Day 43, and one was withdrawn by the investigator due to protocol violation (positive drug screen on Day 120).
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 31
µg/mL |  | 402 (134)

4. Secondary Outcome: Time to Maximum Observed Plasma Concentration of ETI-204 (Tmax) After a Dose of 16 mg/kg on Day 1(Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: Blood samples were obtained and serum concentrations were determined using a validated enzyme-linked immunosorbent assay method with an assay range of 100 ng/mL to 5000 ng/mL.The PK parameter, Tmax, was derived from ETI-204 serum concentrations by sequence group and treatment period for the PK analysis population. Sequence A - there were insufficient serum concentration data to adequately characterize ETI 204 PK separately after each dose administration (Day 1 and Day 14), therefore it was treated as one 32 mg/kg dose split into two 16 mg/kg administrations. Sequence B was treated as 2 separate 16 mg/kg doses (Day 1 and Day 120). All 70 subjects who received ETI-204 were included in the PK population: 35 in Sequence A and 35 in Sequence B; however, the full complement of PK parameters could not be determined in all subjects.
Time Frame: as for outcome 2
Population: One subject in Sequence A was prematurely discontinued from the study by the investigator afte the 1st dose of ETI-204 because of AEs. This subject did not receive the 2nd dose of ETI-204 on Day 14 and therefore all PK parameters from this subject were excluded from descriptive statistics.
Measure: Median (Full Range); unit: days
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 34 | 35
days | 13.1 [0.125 to 14.0] | 0.125 [0.0625 to 1.00]

5. Secondary Outcome: Time to Maximum Observed Plasma Concentration of ETI-204 (Tmax) After a Dose of 16 mg/kg on Day 120 (Sequence B)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 31
days |  | 0.0743 [0.0618 to 1.00]

6. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-last) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: PK parameters for 1 subject in Sequence A were excluded because the subject was discontinued after the 1st dose of ETI-204 because of AEs and did not receive the 2nd dose. 2 subjects in Sequence A and 1 subject in Sequence B (Day 1) were missing the final 3 or more scheduled samples and therefore AUC and lambda z-based parameters were not reported.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 32 | 34
µg.day/mL | 10,200 (2,500) | 4550 (1220)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-last) After a Dose of 16 mg/kg ETI-204 on Day 120 (Sequence B)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: 4 subjects in Sequence B were excluded because the subjects did not receive the 2nd dose of ETI-204 on Day 120 (1 due to AEs after 1st dose, 1 withdrew consent , 1 lost to follow-up, 1 protocol violation). 1 subjects in Sequence B was missing the final 3 or more scheduled samples and therefore AUC and lambda z-based parameters were not reported.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 30
µg.day/mL |  | 4300 (1010)

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 191 Days (AUC0-191days) After a Dose of 16 mg/kg ETI-204 on Days 1 and 14 (Sequence A)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: PK parameters for 1 subject in Sequence A were excluded because the subject did not rec a 2nd dose of ETI-204 due to AEs after the 1st dose. 2 subjects in Sequence A were missing the final 3 or more scheduled samples and therefore AUC and lambda z-based parameters were not reported. AUC0-191days was not calculated for Sequence B.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 32 | 0
µg.day/mL | 10,300 (2480) |

9. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 120 Days (AUC0-120days) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B)
Description: as for outcome 3
Time Frame: On Day 1 predose, at the end of infusion, and 3 and 8 hours after the start of infusion, and on Days 2, 8, 15, 28, 43, 71, 85, 121, 128, 134, 149, 163, and 191.
Population: One subjects in Sequence B was missing the final 3 or more scheduled samples (subject withdrew from the study on Day 8 due to conflict with work schedule) and therefore AUC and lamda z-based parameters were not reported. AUC0-120days was not calculated for Sequence A.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 34
µg.day/mL |  | 4560 (1220)

10. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: PK parameters for 1 subject in Sequence A were excluded because the subject was discontinued after the 1st dose of ETI-204 because of AEs and did not receive the 2nd dose. 2 subjects in Sequence A and 1 subject in Sequence B were missing the final 3 or more scheduled samples and therefore AUC and lambda z-based parameters were not reported.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 32 | 34
µg.day/mL | 10,300 (2530) | 4690 (1370)

11. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) After a Dose of 16 mg/kg ETI-204 on Day 120 (Sequence B)
Description: as for outcome 3
Time Frame: On Day 120 prepose, at the end of infusion, and 3 and 8 hours after the start of infusion, and on Days 2, 8, 15, 28, 43, 71, 85, 121, 128, 134, 149, 163, and 191.
Population: 4 subjects in Sequence B were excluded because they did not receive the 2nd dose of ETI-204 on Day 120. For 4 subjects in Sequence B the AUC and lambda z-based parameters were excluded from descriptive statistics for Day 120 (1 for missing the final 3 or more scheduled samples, 3 because the t1/2 values were >50% of the sample collection interval).
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 27
µg.day/mL |  | 4400 (796)

12. Secondary Outcome: Terminal Half-life (t1/2) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 32 | 34
days | 22.8 (5.82) | 21.5 (6.73)

13. Secondary Outcome: Terminal Half-life (t1/2) After a Dose of 16 mg/kg ETI-204 on Day 120 (Sequence B)
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 27
days |  | 18.6 (3.43)

14. Secondary Outcome: Systemic Clearance (CL) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: PK parameters for 1 subject in Sequence A were excluded because the subject was discontinued after the1st dose of ETI-204 because of AEs and did not receive the 2nd dose. 2 subjects in Sequence A and 1 subject in Sequence B were missing the final 3 or more scheduled samples and therefore AUC and lambda z-based parameters were not reported.
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 32 | 34
Liters/day | 0.274 (0.0862) | 0.300 (0.104)

15. Secondary Outcome: Systemic Clearance (CL) After a Dose of 16 mg/kg ETI-204 on Day 120 (Sequence B)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 27
Liters/day |  | 0.313 (0.0760)

16. Secondary Outcome: Volume of Distribution (Vd) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B) or Two Doses on Days 1 and 14 (Sequence A)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 32 | 34
Liters | 8.69 (2.65) | 8.75 (2.09)

17. Secondary Outcome: Volume of Distribution (Vd) After a Dose of 16 mg/kg ETI-204 on Day 120 (Sequence B)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 27
Liters |  | 8.33 (2.39)

18. Secondary Outcome: Volume of Distribution at Steady State (Vdss) After a Dose of 16 mg/kg ETI-204 on Day 1 (Sequence B)
Description: as for outcome 3
Time Frame: as for outcome 9
Population: One subject in Sequence B was missing the final 3 or more scheduled samples and therefore AUC and lambda z-based parameters were not reported. Vdss was not reported for Sequence A.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 34
Liters |  | 7.20 (1.49)

19. Secondary Outcome: Volume of Distribution at Steady State (Vdss) After a Dose of 16 mg/kg ETI-204 on Day 120 (Sequence B)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 27
Liters |  | 7.01 (2.32)

20. Secondary Outcome: Number of Participants With Anti-ETI-204 Antibodies
Description: Serum anti-ETI-204 antibody titers were determined for all subjects in the safety population. Blood samples were collected and serum samples were assayed at an initial dilution of 1:10. Samples that were positive at the 1:10 dilution were serially diluted 1:2 and assayed until a negative result was attained. The titer of the most dilute sample yielding a positive result was recorded as the titer for that time point. Immunogenicity was measured by the number of participants in each study arm with anti-ETI-204 antibody values post-treatment ≥ 4-times higher than baseline at Day 8, 43 or 71, or if the titer was negative at baseline, the post-treatment sample(s) required a titer of at least 1:20 for it to be considered positive.
Time Frame: On Days 1,14, and 120 predose and on Days 8, 43, 85, 128, 163, and 191
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 35 | 35
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 191 days or 221 days (30 days after the final study visit) for subjects with ongoing adverse events at the final study visit, for each arm
Arm/Group | Sequence A | Sequence B
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35
Other Adverse Events (participants affected / at risk) | 30/35 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence A (N=35) | Sequence B (N=35)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — One subject experienced an ankle fracture on Day 166 and was hospitalized. This event was considered not related to the study drug by the investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence A (N=35) | Sequence B (N=35)
Somnolence (Nervous system disorders) | 10 (19) | 10 (16)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 11 (11)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (6)
Infusion site swelling (General disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 3 (4) | 3 (3)
Infusion site erythema (General disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Infusion site pain (General disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Phlebitis superficial (Vascular disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the sponsor and are confidential. Written approval from the sponsor is required prior to disclosing any information related to this clinical study.